CLINICAL TRIAL: NCT02843555
Title: The Etiology, Pathogenesis, and Natural History of the Leukodystrophies
Brief Title: Natural History of the Leukodystrophies
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 008-169
Record Dates: First submitted 2016-04-07; First posted 2016-07-26 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Leukodystrophies
Keywords: Leukodystrophy; Myelin Gene; Myelin Protein; Sural Nerve Biopsy; Undiagnosed Disease; Schwann Cell; White Matter Pathology; Motor Delay; Cognitive Regression; Motor Deterioration; Unknown Disease
MeSH Terms: conditions — Undiagnosed Diseases; Psychomotor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, skin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Leukodystrophy of unknown etiology: Subjects who may have an undiagnosed form of leukodystrophy

SUMMARY:
The purpose of this study is to:

1. define novel homogeneous groups of patients with LDs and
2. work toward finding the cause of these disorders.

DETAILED DESCRIPTION:
Patients with leukodystrophies (LDs) of unknown etiology are a heterogeneous group but constitute the second largest group of genetic white matter diseases. In order to find the cause of leukodystrophies, patients with LDs of unknown cause will be analyzed clinically, neurophysiologically, biochemically and genetically. Patients would have been diagnosed as having no known leukodystrophies at outside centers. At the Baylor University Medical Center, such patients will undergo a series of neuropsychological, blood, urine, spinal fluid, radiological, and peripheral tissue pathological tests. Some of these tests will be part of a standard battery while others will be tailored to individual patients. Patients will be followed yearly or as necessary. Patients will be screened for mutations in genes coding for structural myelin proteins. In some patients in whom all tests yielded no information regarding the etiology of their disease, and in whom there is evidence to suggest involvement of the peripheral nervous system, a sural nerve biopsy will be considered. Sural nerve biopsy tissue will be evaluated using a novel combination of approaches including detailed pathological, immunohistochemical, and biochemical analysis of myelin proteins and lipids. Schwann cell biology and expression of myelin genes in the brain will also be investigated in situ. It is hoped that the present study will help clarify the nosology of the leukodystrophies and significantly advance our understanding of the pathogenesis of these diseases.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* have clinical and radiographic signs of leukodystrophy without a specific etiology
* no diagnosis of adrenoleukodystrophy, adrenomyeloneuropathy, metachromatic leukodystrophy, Krabbe disease, Canavan disease, a well-defined amino acid organic acid disorder, or a systemic mitochondrial cytopathy.
* First-degree relatives of patients with leukodystrophies of unknown etiology (father, mother, siblings, or sons and daughters of the patients)
* Be able to travel to Baylor University Medical Center in Dallas Texas for evaluation and spend 5-8 working days on site
* Be able to tolerate a general exam and neurological exam
* Be able to tolerate a modest amount of blood drawing, provide a urine specimen, and have a skin biopsy(if not previously done)
* Be able to tolerate the performance of necessary neuroimaging studies to include EEG and Head MRI
* Be able to tolerate a neuropsychological testing and rehabilitation evaluation
* Be able to tolerate spinal tap or nerve biopsy if needed

Exclusion Criteria:

* Unable to travel to Baylor University Medical Center in Dallas Texas for evaluation
* Refusal to sign a study consent form
* Unable to tolerate the performance of the required testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects identified with a leukodystrophy of unknown etiology
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Neuropsychological evaluation to measure baseline cognitive function and detect signs of dementia over time | Every 52 weeks up to 5 years
  Neuropsychological status is evaluated at Baseline and no less than once every year for the duration of the study to assess for any deterioration in function

SECONDARY OUTCOMES:
Evoked potentials to assess involvement of different areas of brain over time | Every 52 weeks up to 5 years
  Evoked potentials are evaluated at Baseline and no less than once every year for the duration of the study to assess for changes in function
MRI of the brain to assess involvement of different areas of the brain over time | Every 52 weeks
  Changes in the brain are assessed at Baseline and no less than once every year for the duration of the study to assess for changes
Electroencephalogram to assess involvement of different areas of the brain over time | Every 52 weeks up to 5 years
  EEG is assessed at Baseline and no less than once a year for the duration of the study to assess for changes in function
Electromyelogram to assess for changes in muscle function over time | Every 52 weeks up to 5 years
  EMG is assessed at Baseline and no less than once a year for the duration of the study to assess for changes in function
Nerve Conduction study to assess abnormalities in affected nerves | Every 52 weeks up to 5 years
  Nerve conduction is assessed at Baseline and no less than once a year for the duration of the study to assess for changes in function
Skin biopsy for to look for evidence of storage disease | Baseline
DNA Studies to search for mutations in genes of structural myelin proteins or genes that control myelin production | Baseline
Spinal Tap to look for diagnostic markers of leukodystrophy | Baseline
Nerve Biopsy to look for pathological abnormalities in affected nerves | Baseline
Neuro-ophthalmological exam to assess for abnormalities in the eye | Every 52 weeks up to 5 years
  Eyes are assessed at Baseline and no less than once a year for the duration of the study to assess for changes in function

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Schiffmann, MD, MHS, Principal Investigator — Baylor University Medical Center, Baylor Institute of Metabolic Disease
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No